CLINICAL TRIAL: NCT04126447
Title: Platelet Indices ( Platelet Count - Mean Platelet Volume - Platelet Distribution Width ) in Decompensated Post Hepatitic Liver Cirrhosis
Brief Title: Platelet Indices in Decompensated Post Hepatitic Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Nader Asham, principle investigator, Assiut University
Other Study IDs: Platelet in cirrosis
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: MPV; PDW

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present work is to study platelet indices ( platelet count - mean platelet volume - platelet distribution width ) as noninvasive predictors in decompensated post hepatitic liver cirrhosis .

DETAILED DESCRIPTION:
Cirrhosis is an advanced liver disease characterized by fibrosis and alteration in hepatic architecture with the development of structurally anomalous nodules . Ascites is a condition in which pathological collection of fluid occurs within the peritoneal cavity mainly because of portal hypertension. It is a major complication of liver cirrhosis, The appearance of ascites in cirrhotic patients indicates a poor prognosis , Spontaneous bacterial peritonitis is a severe infection, commonly occurring in cirrhotic ascitic patients.

Platelets are attributed to preserve hemostasis. Yet, recently, there has been growing recognition that they also play an essential role in inflammatory and immune response. Platelets release prothrombotic and proinflammatory agents and participate in the induction and advancement of vascular and inflammatory disorders . Larger-sized platelets contain many granules, and are therefore more efficient in their hemostatic and proinflammatory actions . This is why the mean platelet volume (MPV) and platelet distribution width (PDW) are worth considering as potential tests for platelet function and activation .

The MPV and PWD can be calculated using almost all automated hematology analyzers. The MPV indicates the average platelet size in femtoliters. The PDW, reflecting homogeneity of platelet size, is calculated from the MPV by the equation (SD of platelet volume divided by MPV×100) or the distribution width at 20% frequency .

ELIGIBILITY:
Inclusion Criteria:

* post hepatitic liver cirrhotic patients

Exclusion Criteria:

* renal failure patients
* pregnents
* diabetic patients
* patients with bone marrow disorders specially platelet disorders
* patient with other cause of liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of the present work is to study platelet indices as noninvasive predictors in decompensated post hepatitic liver cirrhosis .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
platelet indices ( platelet count - mean platelet volume - platelet distribution width ) in decompensated post hepatitic liver cirrhosis | 3 years
  The aim of the present work is to study platelet indices ( platelet count - mean platelet volume - platelet distribution width ) as noninvasive predictors in decompensated post hepatitic liver cirrhosis .